CLINICAL TRIAL: NCT06053879
Title: Biofeedback Intervention in Rehabilitation of Adolescence With Posterior Sagittal Anorectoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Noha Ahmed Fouad Abd-Elrahman, lecturer of physical therapy for women health, Badr University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BUC-IACUC-230507-20
Record Dates: First submitted 2023-09-11; First posted 2023-09-26 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Fecal Incontinence in Children
MeSH Terms: interventions — Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: pretest post test
Masking Description: biofeedback stimulation for faecal incontinence post Posterior Sagittal Anorectoplasty
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biofeedback electrical stimulation (Experimental): Biofeedback electrical stimulation
  Interventions: Other: Biofeedback electrical stimulation

INTERVENTIONS:
Other: Biofeedback electrical stimulation — biofeedback stimulation for faecal incontinence post Posterior Sagittal Anorectoplasty
  Other Names: Biofeedback

SUMMARY:
most of children undergo Posterior Sagittal Anorectoplasty Complain from faecal incontinence and faecal soiling which negatively impacts the social life of these children prohibiting their participation with their bears.

DETAILED DESCRIPTION:
most of children undergo Posterior Sagittal Anorectoplasty Complain from faecal incontinence and faecal soiling which negatively impacts the social life of these children prohibiting their participation with their bears so this study aims prevent faecal incontinence so continue life time without any interference with social life and activities

ELIGIBILITY:
Inclusion Criteria:

* Age from 10-13 years old
* Reliable females
* Able to understand verbal commands
* Normal vision and hearing

Exclusion Criteria:

* Neuromuscular or musculoskeletal disorders
* Behavioural disorders
* Psychological disorders

Ages: 10 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
EMG biofeedback assessment for contraction of anus and puborectalis muscle | 12 weeks
  EMG biofeedback assessment for degree ofanal contraction in cases with faecal incontinence post Posterior Sagittal Anorectoplasty

CONTACTS AND LOCATIONS:
Overall Officials: Reham A Elkalla, PHD, Principal Investigator — Lecturer of PT for surgery and burn; Mostafa S Ali, PHD, Principal Investigator — Ass.Prof. of PT for paediatric; Radwa S Mahmoud, PHD, Principal Investigator — Ass.Prof. of PT for paediatric; Noha A Abd el rahman, PHD, Principal Investigator — lecturer of PT for women health
Locations (1):
- Badr university in cairo, Badr, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No